CLINICAL TRIAL: NCT06574919
Title: Clinical and Functional Assessment of Patients With Inherited Non-Duchenne Myopathies in Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Nasser Abdelaal, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-24-07-15MS
Record Dates: First submitted 2024-08-12; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Inherited Non-Duchenne Myopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases group: patients with inherited non-Duchenne Myopathies

SUMMARY:
Muscular Myopathies are a heterogenous group of inherited muscular disorders characterized by progressive muscle weakness. Historically, these disorders are difficult to treat. In the last three decades, there is a great progress in molecular and genetic basis of these disorders; early diagnosis is achievable with proper clinical recognition and advanced genetic testing [1].

Duchenne Muscular Dystrophy (DMD) is a neuromuscular muscular X-linked recessive disorders that belong to a group of disorders known as dystrophinopathies. DMD is caused by mutations in the dystrophin gene that placed in the middle of short arm of X chromosome [2]. Mutation in this gene lead to absence of dystrophin or structural defects of this protein. The lack of functional dystrophin impairs the structure and function of myofibers which are essential for physiological growth of muscle tissue [3].

The non-dystrophic myopathies are a group of inherited myopathies defined by distinctive static histochemical and/or characteristic ultrastructural changes on muscle.

The nomenclature of dystrophic myopathies can be confusing as some of them are classified by age of onset of symptoms (e.g., congenital muscular dystrophies), whereas others are classified by distribution of weakness (e.g., limb-girdle muscular dystrophies, distal myopathies, facioscapulohumeral dystrophy, and oculopharyngeal muscular dystrophy), by characteristic clinical features (e.g., myotonic dystrophy), by the name of the causative gene (e.g., GNE-myopathy, dystrophinopathies), whereas others are named after the physician first describing the disease (i.e., Duchenne and Becker muscular dystrophy or Bethlem myopathy) or can be subdivided in an entirely different way (i.e., the subgroups of the limb-girdle muscular dystrophies which were named according to their mode of inheritance and order of publication) ]4[ Several aspects need to be taken into account in order to establish a clinical diagnosis; these features include but are not limited to the severity of the muscular wasting, as well as its distribution, and the accompanying symptomology, biochemical, hematological, physical, and neurological investigations, electromyography, and muscle biopsy. Moreover, if the gene defect is established, diagnosis can also be confirmed by gene testing ]5[

Muscle biopsy lacks of typical dystrophic features such as increased conjunctive endomysial tissue, necrosis, and regeneration and shows one or more characteristic histological features. Based in pathological descriptions, the main non-dystrophic myopathies were described during the last century, taking into account the age of onset and the structural or ultrastructural markers [6].

Certain genes, in particular those with large sizes (TTN, RYR1, NEB), may present with different clinical and histological phenotypes and therefore their related myopathies be classified within different groups [7].

It is useful to know that other genetic myopathies may mimic non-dystrophic myopathies. This is the case of certain metabolic and mitochondrial myopathies that may show very selective muscle weakness. The description of these disorders goes beyond the scope of this chapter. However, it may be useful to take into account at least three examples, Pompe disease, the glycogen storage disorder type II (GSD II), and TK2-related mitochondrial DNA depletion myopathy, because they may present as congenital or later-onset non-dystrophic myopathies, may show particular muscle imaging abnormalities, and may be treatable [8; 9].

Understanding the clinical and molecular characteristics of non-DMD is crucial for several reasons. First, accurate diagnosis is essential for proper genetic counseling and family planning. Second, identification of the specific genetic mutation allows for the potential development of targeted therapies in the future. Finally, characterization of the clinical course of different non-DMD can guide treatment decisions and improve patient outcomes.

DETAILED DESCRIPTION:
Type of the study:

This study will be a prospective, observational study

Place of the study:

Pediatric Neurology Clinic and Genetics Unit, Department of pediatrics, Sohag University Hospital. , Sohag, Egypt.

Study duration:

One year (starting from obtaining approval from the research ethics committee).

Study Population:

Children diagnosed with non-DMD at Sohag University Hospital will be included in the study.

Inclusion criteria:

* Age between 2 and 18 years
* Confirmed diagnosis of non-DMD based on clinical features, laboratory investigations, and genetic testing.
* Patients and their parents agree to participate in the study.

Exclusion criteria:

* Children with a confirmed diagnosis of DMD
* Children with incomplete medical records or unavailable clinical data.
* Children with endocrinal ,nutritional critical care and inflammatory myopathies.
* Other neuromuscular disorders that affect AHC or nerves as SMA, congenital myasthenia Gravis and neuropathic.
* Other acquired neuromuscular disorders as Guillain Barre syndrome and toxic myopathy.
* Patients and their parents refuse to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 2 and 18 years

  * Confirmed diagnosis of non-DMD based on clinical features, laboratory investigations, and genetic testing.
  * Patients and their parents agree to participate in the study.

Exclusion Criteria:

* • Children with a confirmed diagnosis of DMD

  * Children with incomplete medical records or unavailable clinical data.
  * Children with endocrinal ,nutritional critical care and inflammatory myopathies.
  * Other neuromuscular disorders that affect AHC or nerves as SMA, congenital myasthenia Gravis and neuropathic.
  * Other acquired neuromuscular disorders as Guillain Barre syndrome and toxic myopathy.
  * Patients and their parents refuse to participate in the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Age between 2 and 18 years
  * Confirmed diagnosis of non-DMD based on clinical features, laboratory investigations, and genetic testing.
  * Patients and their parents agree to participate in the study
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and Functional Assessment of patients with Inherited Non-Duchenne Myopathies in Sohag University Hospital | 1 year
  Characterize the clinical, laboratory, radiological, electrophysiological and molecular features of patients with non-Duchenne muscular dystrophies

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Sohag university Hospital, Sohag
  - Sohag University, Sohag
  - Sohag University Hospital, Sohag

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharawat IK, Ramachandran A, Panda PK, Elwadhi A, Tomar A. Development and Validation of an Outpatient Clinical Predictive Score for the Diagnosis of Duchenne Muscular Dystrophy/Becker Muscular Dystrophy in Children Aged 2-18 Years. Ann Indian Acad Neurol. 2023 Jul-Aug;26(4):453-460. doi: 10.4103/aian.aian_20_23. Epub 2023 Jun 12. PMID 37970286
- [Background] Kim J, Jung IY, Kim SJ, Lee JY, Park SK, Shin HI, Bang MS. A New Functional Scale and Ambulatory Functional Classification of Duchenne Muscular Dystrophy: Scale Development and Preliminary Analyses of Reliability and Validity. Ann Rehabil Med. 2018 Oct;42(5):690-701. doi: 10.5535/arm.2018.42.5.690. Epub 2018 Oct 31. PMID 30404418
- [Background] Lue YJ, Su CY, Yang RC, Su WL, Lu YM, Lin RF, Chen SS. Development and validation of a muscular dystrophy-specific functional rating scale. Clin Rehabil. 2006 Sep;20(9):804-17. doi: 10.1177/0269215506070809. PMID 17005504
- [Result] North KN, Wang CH, Clarke N, Jungbluth H, Vainzof M, Dowling JJ, Amburgey K, Quijano-Roy S, Beggs AH, Sewry C, Laing NG, Bonnemann CG; International Standard of Care Committee for Congenital Myopathies. Approach to the diagnosis of congenital myopathies. Neuromuscul Disord. 2014 Feb;24(2):97-116. doi: 10.1016/j.nmd.2013.11.003. Epub 2013 Nov 18. PMID 24456932